CLINICAL TRIAL: NCT00573105
Title: Laparoscopic Ventral Hernia Repair by Heavy Weight or Lighter Weight Mesh (COMPOSIX-trial)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow inclusion rate
Sponsor: University Hospital, Ghent (Other)
Collaborators: C. R. Bard (Industry)
Responsible Party: Frederik Berrevoet, University Hospital Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/421
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Laparoscopic Ventral hernia repair by heavy weight mesh
  Interventions: Procedure: Laparoscopic Ventral hernia repair by heavy weight mesh
- 2 (Experimental): Laparoscopic Ventral hernia repair by lighter weight mesh
  Interventions: Procedure: Laparoscopic Ventral hernia repair by lighter weight mesh

INTERVENTIONS:
Procedure: Laparoscopic Ventral hernia repair by heavy weight mesh — Laparoscopic Ventral hernia repair by heavy weight mesh
  Arms: 1
Procedure: Laparoscopic Ventral hernia repair by lighter weight mesh — Laparoscopic Ventral hernia repair by lighter weight mesh
  Arms: 2

SUMMARY:
1. General

   - antibiotic prophylaxis: cefazoline (Cefacidal™) 2 gram iv administered 30 minutes before surgery
2. Laparoscopic surgery

   * at least 5 cm overlap (mesh diameter should exceed hernia size by at least 10 cm)
   * with or without anchoring transparietal sutures or double crown technique

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from the patient or his/her legal representative
* ventral hernia requiring elective surgical repair

Exclusion Criteria:

* no written informed consent
* 'hostile' abdomen; open abdomen treatment
* contraindication to pneumoperitoneum
* emergency surgery (incarcerated hernia)
* parastomal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
recurrence rate | after 1 year

SECONDARY OUTCOMES:
morbidity rate | perioperative
quality of life | after 1 year
postoperative pain | within 1 week
long term complication rate | after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be